CLINICAL TRIAL: NCT00694226
Title: Brief Intervention in Substance Use Among Adolescent Psychiatric Patients: A Randomized Controlled Trial
Brief Title: Brief Intervention in Substance Use in Adolescent Psychiatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Josefina Castro-Fornieles / Chief of the Child and Adolescent Psychiatry and Psychology departement, Hospital Clinic Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1719/2003
Record Dates: First submitted 2008-05-23; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Substance-Related Disorders
Keywords: Adolescent; Substance use; Brief intervention; Child psychiatry
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Brief intervention, consisting in an intervention with the adolescent and a session with parents or mentors. The session with the adolescent lasted 60 minutes. Materials related to the interview were developed according to previous reports on the subject. After building a good rapport the interviewer involved the patient in an initial discussion about the results of the evaluation. This led to a review of the drugs used by the subject and an elicitation of positives and negatives of drug use. The relationship between drug use and current and long-term goals was explored. Discrepancies and problems in the future related to substance use were examined, and information and counseling was offered. The basic components of the motivational interview approach were contemplated, and several skills were used by the interviewers. The individual session with parents or mentors consisted in the presentation of educational materials and a brief counseling intervention on parenting skills.
  Interventions: Behavioral: brief motivational intervention
- 2 (Active Comparator): Treatment as usual (TTU): Individuals assigned to this group and their parents or tutors received standard care and no further intervention other than completion of the assessment protocol. After completing the assessment individuals and their families went on to receive standard care at the Child and Adolescent Psychiatry and Psychology Department according to the primary diagnosis
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: brief motivational intervention — Brief intervention, consisting in an intervention with the adolescent and a session with parents or mentors. The session with the adolescent lasted 60 minutes. Materials related to the interview were developed according to previous reports on the subject. After building a good rapport the interviewer involved the patient in an initial discussion about the results of the evaluation. This led to a review of the drugs used by the subject and an elicitation of positives and negatives of drug use. The relationship between drug use and current and long-term goals was explored. Discrepancies and problems in the future related to substance use were examined, and information and counseling was offered. The basic components of the motivational interview approach were contemplated, and several skills were used by the interviewers. The individual session with parents or mentors consisted in the presentation of educational materials and a brief counseling intervention on parenting skills.
  Arms: 1
Behavioral: treatment as usual — Treatment as usual (TTU): After completion of the intervention, individuals and their families went on to receive standard care at the Child and Adolescent Psychiatry and Psychology Department according to the primary diagnosis.Individuals assigned to this group and their parents or tutors received standard care and no further intervention other than completion of the assessment protocol.
  Arms: 2

SUMMARY:
The objective of the study was to assess the efficacy in decreasing the likelihood of substance use of a brief motivational enhancement intervention in adolescents referred to psychiatric treatment.

237 adolescents consecutively admitted to a psychiatry department completed an evaluation of their substance use. Subjects identified as users were randomly allocated to one of two groups: an experimental group that received a brief intervention aimed at increasing their awareness of the risks of substance use, or a control group. All subjects received standard treatment according to the primary diagnosis. Structured questionnaires assessing knowledge, attitudes, perception of risks and intention of use of psychoactive substances were administered upon admission and 1 month later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 12-17
* consecutively referred for psychiatric or psychological assessment and treatment to a Child and Adolescent Psychiatry and Psychology Department

Exclusion Criteria:

* Not willing to take part.
* Mentally retarded
* Non completion of a substantial part of the assessment protocol.
* Presenting severe acute psychopathological disturbances that interfere with the assessment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2004-03; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Attitudes towards psychoactive substances (Knowledge, Risk perception, Problems and Intention of use) measured with questionnaires obtained from the Evaluation Instruments Bank (EIB), European Monitoring Centre for Drugs and Drug Addiction (EMCDDA). | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain